CLINICAL TRIAL: NCT06832501
Title: Effectiveness of the Henna Application in Patients with Hand-Foot Syndrome: Nested Case-Control Study
Acronym: [Henna]
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Berna KURT, Assistant professor, Hacettepe University
Other Study IDs: KA-180085
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Henna; Hand-Foot Syndrome; Case-Control Study
Keywords: Capecitabine; palmar-plantar erythrodysesthesia; symptom management; hand-foot syndrome
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — lawsone; Diagnosis-Related Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Case group/Control group: In the data collection process, 84 patients received capecitabine and two patients (1:2) who met the inclusion criteria served as the control group (n=56, who received the test) for each case (n=28).
  Interventions: Other: Henna

INTERVENTIONS:
Other: Henna — The day-care unit of the University of Hacettepe's oncology hospital is being trained by educational nurses on the treatment of patients receiving capecitabine a day before the application of chemotherapy. All the patients were questioned about their individual and disease-related characteristics using the Patient Information Form, and The National Cancer Institute common terminology criteria for adverse events - version 4.03 (NCICTCAE v4.03), EORTC C30 Cancer Quality of Life Scale, and The Hand-Foot Syndrome-14 (HFS-14) were used by face-to-face interview technique.On the 21st day and the 63rd day after the first treatment course, patients who developed hand-foot syndrome constituted the case-control group, including patients who applied henna and patients who did not apply henna.
  Other Names: case group

SUMMARY:
Introduction: There is an explanation that there is a connection between the application of henna and the occurrence of hand-foot syndrome, and the purpose and progression of this interaction. This nested case-control study of participants who underwent capecitabine therapy were breast and colorectal cancer was carried out to prospectively investigate the relationship of hand-foot syndrome with the henna application.

Method: Nested Case-Control (NCC) design within a longitudinal observational prospective cohort study in the setting of an oncology clinic. The primary outcome was hand-foot syndrome from in-hospital interviews and medical record reviews. In the data collection process, 84 patients received capecitabine and two patients (1:2) who met the inclusion criteria served as the control group (n=56, who received the test) for each case (n=28). The case and control groups were followed for 12 weeks. HFS-14 Scale and EORTC QLQ-C30 Quality of Life were conducted on the baseline, first follow-up (T1=day 21), and second follow-up (T2=day 63) cycles of chemotherapy. We used a non-parametric signed-rank test to test the median of paired differences.

DETAILED DESCRIPTION:
Capecitabine is among the most effective treatments for metastatic or late-stage breast cancer. It is also another treatment approach for colorectal cancer. Capecitabine is a high-concentration 5-FU prodrug planned for thymidine phosphorylase enzyme primarily for two cancer types [1, 2]. Hand-foot syndrome (HFS), increasing skin pigmentation, diarrhea, nausea-vomiting, and fatigue are common side effects of the capecitabine treatment. According to phases 1 and 2 studies, the most common side effect of capecitabine is HFS, with a frequency that ranges from 10 to 50.7% [3]. HFS is a serious condition characterized by the accumulation of symmetrical, sharply contained, erythematous, edematous plaques, particularly on the lateral parts of the fingers, the thenar and hypothenar processes, after a symptomatic period in which scorching occurs. The soreness experienced by the patients limits their daily routines [4], and their quality of life is negatively impacted because of their incapacity to function in their hands and feet.

Hand-foot syndrome has been observed to occur during the second cycle of treatment [5]. There remains no currently effective treatment for this side effect today. Previous case reports indicate that henna may successfully safeguard against and halt the evolution of HFS [6, 7]. Henna (Lawsonia inermis L.) as a plant of the Myrtales order, classified under the Lythraceae family. Henna possesses a 9000-year history and has played a crucial role in herbal treatment since the Ayurvedic era [8]. Henna is a pigment derived from the desiccated bark and leaf of "Lawsonia inermis." Since the Lawsone molecule can combine with proteins, it is frequently used to color nails, the epidermis, hair, and clothing. Henna leaves are powdered, diluted in water or oil to make them stronger, and afterward applied to the skin, penetrating through the upper layer of the skin and turning a dark red color. It is a healthy and without side effects application. The growth and development inhibition of the extract on Candida albicans was identified in studies utilizing water, methanol, and chloroform extraction of henna leaves, and its antifungal activity was explained [9]. Until now, Hosein and Zinab's study revealed that water and methanol extracts of henna plant leaves possessed significant antioxidant qualities [8]. In another investigation that looked at antioxidant activity, the leaves were extracted with various solvents, and it was observed that chloroform extraction constructed the most activity [10].

Among the chemical components of the henna plant, Lawsone (LW), MCF-7, Caco-2, BJ, and Keratinocyte cells were evaluated for their efficacy in healing structurally damaged wounds. Various concentration principles might well be optimum in each cell line; the specificity of the LW compound to skin cells, particularly keratinocytes, is higher. While it can heal the wound in cells within as little as six hours, the utilization of the LW compound in the formulation of wound-treating products has been demonstrated with these results, when the control cell without LW has yet to attain 40% wound healing [11]. Besides that, it has been demonstrated in trials that coverings protected with Lawsone nano compound in the treatment of burns suppressed inflammation in the wound tissue and accelerated healing [10], and it was also reported in another study that it was beneficial in decubitus wounds [12]. As a result of the LW compound's antibacterial activity against Bacillus subtilis bacteria, it has been determined that the LW compound is suitable to be employed as an antibacterial agent in the struggle against this bacteria [13]. When henna was applied to a patient with pancreatic cancer and 2nd-degree hand-foot syndrome, HFS symptoms almost completely healed, and the patient's concerns such as burning, soreness, and incapacity to walk were abolished without dose limitation until the end of the treatment [14]. In another case study, Henna was applied to ten patients with metastatic breast and colon cancer who experienced HFS. Six patients had third-degree HFS before the study started, whereas four patients had second-degree HFS. Comprehensive improvement was noted in four patients with third-degree HFS, regression to first-degree level in two patients, and complete response in four patients with second-degree HFS as a consequence of henna treatment. It was recommended in these case reports to perform more experimental studies with more patients [15].

There is an explanation that there is a connection between the application of henna and the occurrence of hand-foot syndrome, and the purpose and progression of this interaction. The likely human links have not been completely clarified yet. Henna used in literature reviews has been found to have a substantial impact on reducing the occurrence of hand-foot syndrome. Capecitabine-induced HFS diminishes patients' quality of life and increases their need for medical attention. Patients who struggle to cope with their regular activities (feeding, personal hygiene, etc.) suffer from severe lesions on their feet and hands and may become dependent on others until the symptoms regress or subside. The need for effective treatments to avoid or decrease these symptoms reported in patients is mentioned in the literature [6-13] as much as possible. Although it has been determined that the majority of patients who received capecitabine were using henna as a protective against hand-foot syndrome according to the reports of nurses and researchers in chemotherapy clinics, our study aims to determine whether henna affects the symptoms. This nested case-control study (NCC) involving those receiving capecitabine treatment for breast and colorectal cancer was conducted to comprehensively examine the association between hand-foot syndrome and henna application. The NCC methodology in a prospective cohort research study is used when outcome data are accessible for all participants, although the exposure of interest has not been collected and is challenging or excessively costly to acquire for all patients. An NCC analysis employing comprehensive matching methods provides estimates that are equally efficient and unbiased as those derived from a complete cohort study. NCC with a reduced sample size is not only affordable but also less computationally intensive than analyzing the entire cohort study. If the matching technique has been performed correctly and the selected controls accurately represent those in the cohort research, then the Nested Case-Control (NCC) design has minimal loss of efficiency comparative to the full cohort analysis [16]. The NCC may provide superior validity compared to the whole cohort study due to its matching approach, which improves the adjustment for both measured and unmeasured factors.

ELIGIBILITY:
Inclusion Criteria:

* Would be getting capecitabine as chemotherapy,
* Were aged between 18 and 65,
* Had a diagnosis of either breast or cancer of the colorectal
* Were willing to communicate, literate, and were informed about their diagnosis,
* Were not using psychotropic drugs, anxiolytic, antidepressant, analgesic, or sedative medications,
* Did not have any type of neurological condition or neuropathy, and vi. consented to participate in the study voluntarily.

Exclusion Criteria:

* Were undergoing radiation,
* Were taking supplements such as vitamin E,
* Had previously had capecitabine treatment,
* Had damage to the skin on their hands or feet,
* Were unwilling to voluntarily engage in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the data collection process, 28 patients received capecitabine treatment at the Hacettepe University Hospital of Oncology meeting the research criteria and two patients (n=56, who received the test) who met the inclusion criteria served as the control group for each case. (1:2). Controls were matched with patients in a ratio of two to one depending on age at collection of samples (+3), gender, body surface area index, and skin type data. Minimum number of samples achieved under at least 5% type error and at least 95% power condition. The study used the initial non-development of EAS as a criterion for the HFS scale score, which was studied between "grade 0" and "grade 3" according to the NIC-CTCAE criteria, and was between 18 and 65 years of age.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of Interventions on Outcomes in the HFS Scores | From enrollment to the end of treatment at 63 days
  Hand and foot symptoms scores were measured at the Baseline (T0), T1, and T2.

SECONDARY OUTCOMES:
Effect of Interventions on Outcomes in the EORTC QLQ-C30 Scores | From enrollment to the end of treatment at 63 days
  The case group and control group assessed the subdimension scores of the EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Kurt, Assistant professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Adnan Saygun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Ngo LH, Inouye SK, Jones RN, Travison TG, Libermann TA, Dillon ST, Kuchel GA, Vasunilashorn SM, Alsop DC, Marcantonio ER. Methodologic considerations in the design and analysis of nested case-control studies: association between cytokines and postoperative delirium. BMC Med Res Methodol. 2017 Jun 6;17(1):88. doi: 10.1186/s12874-017-0359-8. PMID 28587598
- [Background] Yucel I, Guzin G. Topical henna for capecitabine induced hand-foot syndrome. Invest New Drugs. 2008 Apr;26(2):189-92. doi: 10.1007/s10637-007-9082-3. Epub 2007 Sep 21. PMID 17885735
- [Background] Ilyas S, Wasif K, Saif MW. Topical henna ameliorated capecitabine-induced hand-foot syndrome. Cutan Ocul Toxicol. 2014 Sep;33(3):253-5. doi: 10.3109/15569527.2013.832280. Epub 2013 Sep 11. PMID 24021017
- [Background] Habbal O, Hasson SS, El-Hag AH, Al-Mahrooqi Z, Al-Hashmi N, Al-Bimani Z, Al-Balushi MS, Al-Jabri AA. Antibacterial activity of Lawsonia inermis Linn (Henna) against Pseudomonas aeruginosa. Asian Pac J Trop Biomed. 2011 Jun;1(3):173-6. doi: 10.1016/S2221-1691(11)60021-X. PMID 23569753
- [Background] Hekmatpou D, Ahmadian F, Eghbali M, Farsaei S. Henna ( Lawsonia inermis) as an Inexpensive Method to Prevent Decubitus Ulcers in Critical Care Units: A Randomized Clinical Trial. J Evid Based Integr Med. 2018 Jan-Dec;23:2515690X18772807. doi: 10.1177/2515690X18772807. PMID 29756474
- [Background] A. Y. Kilcar, B. Cekic, F. Z. B. Muftuler, et al. ''In vitro evaluation of radiolabeled (125 I) methanol extracts of yarrow in cell lines of MCF-7, PC-3, A-549 and Caco-2,'' Journal of Radioanalytical and Nuclear Chemistry 295, no. 1 (2013): 593-599.
- [Background] Hadisi Z, Nourmohammadi J, Nassiri SM. The antibacterial and anti-inflammatory investigation of Lawsonia Inermis-gelatin-starch nano-fibrous dressing in burn wound. Int J Biol Macromol. 2018 Feb;107(Pt B):2008-2019. doi: 10.1016/j.ijbiomac.2017.10.061. Epub 2017 Oct 13. PMID 29037870
- [Background] M. A. Saadabi, ''Evaluation of Lawsonia inermis Linn.(Sudanese henna) leaf extracts as an antimicrobial agent,'' Research Journal of Biological Sciences 2, no. 4 (2007): 419-423.
- [Background] H. K. M. Hosein, D. Zinab, ''Phenolic compounds and antioxidant activity of henna leaf extracts (Lawsonia inermis),'' World Journal of Dairy & Food Sciences 2, no. 1 (2007): 38-41.
- [Background] E. Karimi, B. Gharib, N. Rostami, L. Navidpour, and M. Afshar, ''Clinical efficacy of a topical polyherbal formulation in the management of fluorouracil-associated hand-foot syndrome,'' Journal of Herbal Medicine 17, (2019): 100270.
- [Background] Pandy JGP, Franco PIG, Li RK. Prophylactic strategies for hand-foot syndrome/skin reaction associated with systemic cancer treatment: a meta-analysis of randomized controlled trials. Support Care Cancer. 2022 Nov;30(11):8655-8666. doi: 10.1007/s00520-022-07175-3. Epub 2022 Jun 2. PMID 35655045
- [Background] Jiang Z, Yang Y, Li L, Yue Z, Lan L, Pan Z. Capecitabine monotherapy in advanced breast cancer resistant to anthracycline and taxane: A meta-analysis. J Cancer Res Ther. 2018 Dec;14(Supplement):S957-S963. doi: 10.4103/0973-1482.187384. PMID 30539829
- [Background] Scontre VA, Martins JC, de Melo Sette CV, Mutti H, Cubero D, Fonseca F, Del Giglio A. Curcuma longa (Turmeric) for Prevention of Capecitabine-Induced Hand-Foot Syndrome: A Pilot Study. J Diet Suppl. 2018 Sep 3;15(5):606-612. doi: 10.1080/19390211.2017.1366387. Epub 2017 Nov 2. PMID 29095653
- [Background] Basch E, Dueck AC, Rogak LJ, Mitchell SA, Minasian LM, Denicoff AM, Wind JK, Shaw MC, Heon N, Shi Q, Ginos B, Nelson GD, Meyers JP, Chang GJ, Mamon HJ, Weiser MR, Kolevska T, Reeve BB, Bruner DW, Schrag D. Feasibility of Implementing the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events in a Multicenter Trial: NCCTG N1048. J Clin Oncol. 2018 Sep 11;36(31):JCO2018788620. doi: 10.1200/JCO.2018.78.8620. Online ahead of print. PMID 30204536
- [Background] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Background] A. R. Elif, K. T. Yucel, A. B. Ekincioglu, and I. Gullu, ''Capecitabine induced hand-foot syndrome: a systematic review of case reports,'' Clinical and Experimental Health Sciences 9, no. 2 (2019): 178-91.